CLINICAL TRIAL: NCT03548194
Title: A Phase II Randomised, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of BNC210 in Hospitalised Elderly Patients With Agitation
Brief Title: A Study of BNC210 in Elderly Patients With Agitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bionomics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNC210.008
Record Dates: First submitted 2018-03-27; First posted 2018-06-07 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Agitation in the Elderly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BNC210 (Experimental): Administered orally b.i.d. for 5 days.
  Interventions: Drug: BNC210
- Placebo (Placebo Comparator): Administered orally b.i.d. for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BNC210 — BNC210 300 mg b.i.d
  Arms: BNC210
Drug: Placebo — Placebo b.i.d.
  Arms: Placebo

SUMMARY:
This is a Phase II randomised, double-blind, placebo-controlled study assessing the effects of BNC210 on agitation in hospitalised elderly patients as measured by the Pittsburgh Agitation Scale (PAS). Safety and tolerability of BNC210 will also be assessed.

The secondary objectives of the study include evaluation of the effects of BNC210 on global function in patients with agitation as assessed by the Clinical Global Impression Scale (CGI-S/I).

Participants will receive 5 days of blinded treatment followed by 2 days of follow up.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female elderly patient admitted to hospital and under the care of a specialist Geriatrician
* Determined to have agitation requiring intervention in addition to standard of care behavioural management, as assessed by the Investigator or delegate, after at least 24 hours following admission to hospital.

Key Exclusion Criteria:

* Severe Alzheimer's Dementia (stage 7) as assessed by the Functional Assessment Staging Test (FAST).
* Diagnosed with Severe Parkinson's Disease.
* Premorbid psychotic illness as assessed by the Investigator.
* Evidence of severe organ dysfunction
* Confirmed metastatic malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Absolute change in agitation, as measured by the Pittsburgh Agitation Scale (PAS). | 5 days

SECONDARY OUTCOMES:
Absolute change in global function, as measured by the Clinical Global Impression Scale - Severity and Improvement (CGI-S/I) | 5 days
Proportion of participants reaching the "Non-Agitated" state | 5 days
Time to first reach a "Non-Agitated" state. | 5 days

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Prince of Wales Hospital, Sydney, New South Wales
  - Modbury Hospital, Adelaide, South Australia
  - Northern Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Western Health, Melbourne, Victoria